CLINICAL TRIAL: NCT00536250
Title: Study to Investigate the Pathophysiology of Type 2 Diabetes in Youth
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0102012241; R01HD040787 (NIH)
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Impaired Glucose Tolerance; Pre-diabetes; Childhood Obesity; Insulin Resistance; Metabolic Syndrome
Keywords: Pre-Diabetes; Childhood Obesity; Metabolic Syndrome; insulin resistance; Impaired Glucose Tolerance; Non Alcoholic Fatty Liver Disease; High Molecular Weight Adiponectin; Hypoadiponectinemia
MeSH Terms: conditions — Glucose Intolerance; Pediatric Obesity; Insulin Resistance; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Hypoadiponectinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to determine the role of beta-cell function and insulin resistance in the development of impaired glucose tolerance (IGT) and type 2 diabetes in children and adolescents who have an increased risk of developing type 2 diabetes due to overweight/obesity or a family history of overweight/obesity, diabetes and/or impaired fasting glucose. It is hypothesized that: 1)Obese adolescents with IGT will be more insulin resistant than obese adolescents with NGT. Insulin resistance will be the best predictor of changes in glucose tolerance status., 2)Beta cell function will be impaired in obese adolescents with IGT compared to obese adolescents with NGT., 3)Obese adolescents with IGT will present with greater intramyocellular, intrahepatic and visceral fat than obese adolescents with NGT. Furthermore, obese adolescents with IGT will have larger adipocytes, while having significantly fewer adipocytes compared to obese adolescents with NGT. Obese adolescents with IGT will also have altered expression of key genes related to insulin resistance., and 4)Abnormalities in endothelial function as manifested by low FMD and PAT are already present in obese adolescents with IGT and are linked to insulin resistance.

DETAILED DESCRIPTION:
Type 2 diabetes is a serious and common chronic disease affecting an estimated 6.6% of the U.S. population 20 to 74 years of age. Among children, type 2 diabetes has previously been reported to account for 2% to 3% of all patients with diabetes mellitus. Recent studies, however, indicate that the prevalence of this disorder is increasing in the pediatric population. This phenomenon parallels the increased prevalence of obesity in children and adolescents, particularly in African-American and Hispanic ethnic groups. Despite the wealth of knowledge concerning the epidemiology, pathophysiology and treatment of type 2 diabetes in adults, we know little about the disease in children.Paralleling the rise in childhood obesity and type 2 diabetes is an increase in the metabolic syndrome in youth. The metabolic syndrome, also known as "Syndrome X," is characterized by hypertension, type 2 diabetes, dyslipidemia and obesity. This syndrome was first described in 1966 by Camus and again by Reaven in 1988. Cook et al. showed that the metabolic syndrome is already present in 6.8% of 12-19 year-olds with a BMI between the 85th and 95th percentiles, and in 28.7% of those with a BMI greater than the 95th percentile. In addition, recent studies from our group suggest that risk factors for type 2 diabetes and the metabolic syndrome are already present in overweight children and adolescents. As the degree of obesity worsens, the prevalence of these risk factors greatly increase.Overweight and obese adolescents with NGT and with IGT will be recruited. Progression from NGT to IGT and from IGT to type 2 diabetes will be assessed by annual oral glucose tolerance tests (OGTT). Comprehensive metabolic assessments will be employed to examine within and between group differences in insulin action and beta-cell function at baseline and during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Lean (not overweight or obese) will be defined as a body mass index (BMI) (kg/m2) less than the 85th percentile specific for age and gender, overweight will be defined as a BMI between the 85th and 95th percentiles, and obesity will be defined as a BMI greater than the 95th percentile1. Following the oral glucose tolerance test (OGTT, 75 gm) (HIC #11190), children will be classified as normal glucose tolerant if plasma glucose at two hours is <140 mg/dl and as impaired glucose tolerant if plasma glucose is ≥140 mg/dl. To enter the study all children and adults must be in good general health, have a normal medical history and physical exam, and have no endocrinopathies (normal thyroid function test) or other diseases that might affect glucose metabolism.
* Eligibility will be determined by a comprehensive family and medical history and physical examination prior to enrollment in the study. Tanner stage of pubic breast and gonadal development will be determined by physical examination and by measurements of estradiol, testosterone and IGF1 as biochemical markers of pubertal development.

Exclusion Criteria:

* Medications that are known to alter glucose or insulin metabolism, such as oral steroids, or certain psychiatric medications, such as Celexa, Lithium and Paxil. Children and adults will be excluded from participating in the PAT test if they have a latex allergy. Lean subjects must have at least one parent, grandparent or sibling with overweight/obesity (BMI >25), type 2 diabetes, and/or impaired fasting glucose (IFG) (fasting glucose >100 mg/dl). A fasting plasma glucose level will be obtained via finger stick in parents of potential volunteers in whom status of diabetes or IFG is unknown. Exclusion criteria also include known diabetes or taking any medication that alters liver function and blood pressure. Youth on chronic anti-inflammatory medications or who consume alcohol are also excluded.

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and Adolscents seen at the Yale Pediatric Obesity Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2001-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
glucose tolerance | baseline and follow up
  glucose tolerance status as determined by oral glucose tolerance test - fasting and 2 hour glucoses
insulin resistance | baseline and follow up
  insulin resistance as measured during oral glucose tolerance test by WBISI
hepatic fat content and abdominal fat ratio | baseline and follow up
  hepatic fat content and abdominal fat ratio measured by liver mri and abdominal mri

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, M.D., Principal Investigator — Yale University
Locations (1):
- 47 College Street, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berry D, Savoye M, Melkus G, Grey M. An intervention for multiethnic obese parents and overweight children. Appl Nurs Res. 2007 May;20(2):63-71. doi: 10.1016/j.apnr.2006.01.007. PMID 17481469
- [Result] McCartney CR, Blank SK, Prendergast KA, Chhabra S, Eagleson CA, Helm KD, Yoo R, Chang RJ, Foster CM, Caprio S, Marshall JC. Obesity and sex steroid changes across puberty: evidence for marked hyperandrogenemia in pre- and early pubertal obese girls. J Clin Endocrinol Metab. 2007 Feb;92(2):430-6. doi: 10.1210/jc.2006-2002. Epub 2006 Nov 21. PMID 17118995
- [Derived] Halloun R, Galderisi A, Caprio S, Weiss R. Adipose Tissue Insulin Resistance Is Not Associated With Changes in the Degree of Obesity in Children and Adolescents. J Clin Endocrinol Metab. 2023 Apr 13;108(5):1053-1060. doi: 10.1210/clinem/dgac700. PMID 36469736
- [Derived] Trico D, Prinsen H, Giannini C, de Graaf R, Juchem C, Li F, Caprio S, Santoro N, Herzog RI. Elevated alpha-Hydroxybutyrate and Branched-Chain Amino Acid Levels Predict Deterioration of Glycemic Control in Adolescents. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2473-2481. doi: 10.1210/jc.2017-00475. PMID 28482070
- [Derived] D'Adamo E, Northrup V, Weiss R, Santoro N, Pierpont B, Savoye M, O'Malley G, Caprio S. Ethnic differences in lipoprotein subclasses in obese adolescents: importance of liver and intraabdominal fat accretion. Am J Clin Nutr. 2010 Sep;92(3):500-8. doi: 10.3945/ajcn.2010.29270. Epub 2010 Jun 23. PMID 20573788